CLINICAL TRIAL: NCT02403297
Title: Rapid Point-of-Care Salivary Diagnostic for Periodontal Health
Status: Terminated | Type: Observational
Sponsor: Innovative Diagnostics Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013-1R43DE024015-01
Record Dates: First submitted 2015-03-23; First posted 2015-03-31 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Gingivitis; Periodontal Disease
Keywords: Bleeding gums; Gum inflammation; Saliva
MeSH Terms: conditions — Gingivitis; Periodontal Diseases; Gingival Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 5ml of saliva will be collected. A small sample of the saliva will be used chair side to analyze on the device. The remaining saliva will be aliquoted into five samples and kept frozen until analyzed on a Luminex machine.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy: Saliva will be collected from 58 subjects determined to be "healthy" according to the protocol.
  Interventions: Device: Quik Check PD
- Gingivitis: Saliva will be collected from 58 subjects determined to have gingivitis according to the protocol.
  Interventions: Device: Quik Check PD
- Periodontal disease: Saliva will be collected from 58 subjects determined to have periodontal disease according to the protocol.
  Interventions: Device: Quik Check PD

INTERVENTIONS:
Device: Quik Check PD — The device is not an intervention. It is a device to determine if MMP-8 is present in a subjects saliva.

SUMMARY:
The purpose of this study is to learn if a chair-side testing device will accurately measure levels of a salivary biomarker and thus indicate if a patient has periodontal health, gingivitis or periodontal disease.

DETAILED DESCRIPTION:
Human subjects will participate in this cross-sectional study by attending a single visit where their mouth will be examined and saliva will be collected to help determine the accuracy of a POC salivary diagnostic device. The study population will consist of 174 persons (58 that are orally healthy and have no oral discomfort; 58 that have gingivitis; and 58 that have periodontitis. The device results (i.e., visual and optical scans) will be compared against the Luminex results by two methods: 1) the Bland-Altman procedure and 2) discriminant analysis that examines whether the concentration would correctly identify the subject as health or disease using a defined threshold for MMP-8 levels.

Three groups of individuals will be recruited: those that are orally healthy and do not have any oral discomfort (N=58), those who have gingivitis (i.e., bleeding gums; N=58), and those who have periodontal disease (N=58). The groups will be matched by gender and smoking status. Women are predicted to account for 50% of the participants. The age distribution will be 18 to 95 years. Subjects will not be excluded based on race, gender, or ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of all racial and ethnic groups over 18 years of age;
* At least 20 erupted teeth and the ability to provide expectorated saliva;
* Able and willing to comply with study requirements; and
* Have full understanding of all elements of, and signature and dating of the written informed consent prior to the initiation of protocol specified procedures

Exclusion Criteria:

* Prisoners or institutionalized individuals;
* Persons with acute illness or infectious disease (as evidenced by fever, malaise, sore throat, recurrent cough, lymphadenopathy, swelling and/or a physician consultation);
* Evidence of oral mucosal lesion or ulceration; or
* Use of glucocorticoids or cyclooxygenase inhibitors (i.e. such as ibuprofen, Naprosyn(Aleve) or non-steroidal anti-inflammatory drug) daily for the past two weeks.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three groups of individuals will be recruited: those that are orally healthy and do not have any oral discomfort (N=58), those who have gingivitis (i.e., bleeding gums; N=58), and those who have periodontal disease (N=58). The groups will be matched by gender and smoking status. Women are predicted to account for 50% of the participants. The age distribution will be 18 to 95 years. Subjects will not be excluded based on race, gender, or ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Presence of MMP-8 in the subjects saliva using the Quik Check PD device | One day. Subjects complete the study in 45 minutes.

SECONDARY OUTCOMES:
Amount of MMP-8 in the subjects saliva sample using Luminex Analysis | One day. Subjects complete the study in 45 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Innovative Diagnostics Inc, Lexington, Kentucky, United States